CLINICAL TRIAL: NCT04804137
Title: Immune Response Under Immunotherapy in Metastatic Non-Small Cell Lung Cancer: Sputum, Blood Samples and Microbiota Study
Brief Title: Immune Response Under Immunotherapy in Metastatic NSCLC: Sputum, Blood Samples and Microbioata Study
Acronym: RICEPS
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Collaborators: Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI20-RICEPS
Record Dates: First submitted 2021-03-08; First posted 2021-03-18 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Non-squamous Lung Cancer; Metastatic Lung Cancer
Keywords: Blood sample; sputum; microbiota; Immunotherapy; saliva
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Specimen Collection; Defecation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample, stool, saliva, sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group: adult patients with adenocarcinoma type non-small cell lung cancer
  Interventions: Other: Blood; Other: sputum; Other: saliva; Other: stool

INTERVENTIONS:
Other: Blood — Blood samples are taken at each visit to the day hospital for a programmed injection of immunotherapy.
Other: sputum — induced by saline aerosol sputum during each visit to the day hospital for a programmed injection of immunotherapy.
Other: saliva — spontaneous saliva during each visit to the day hospital for a programmed injection of immunotherapy.
Other: stool — Stool analyses will be carried out on a sample taken by the patient at home and brought back at the time of a day hospital.

SUMMARY:
Prospective pathophysiological exploratory monocentric study, focusing on adult patients with non-small cell lung cancer (NSCLC) : non-squamous type without oncogenic addiction, metastatic, treated with immune checkpoint inhibitors alone or in combination with chemotherapy in front line at the CHRU de Tours, France.

DETAILED DESCRIPTION:
The percentage of patients benefiting from immunotherapy is quite low and their systemic side effects can sometimes be severe. One of the main difficulties is to identify before treatment patients who will respond to immune checkpoint inhibitors. Currently, the selection is done in a very large majority of cases on the expression of PD-L1 by the tumor. But this biomarker is not sufficient to identify patients responding or not to immune checkpoint inhibitors. In addition, factors extrinsic to the tumor, to its microenvironment and patient immunity may be involved in the response to immunotherapy such as the microbiota.

The investigators therefore assume that the immune response in place during immunotherapy treatment differs according to the profile of patient response to immunotherapy.

The main objective of this project is to describe local and systemic anti-tumor immune system of patients responders or not to immune checkpoint inhibitors, but also whether the immunological characterization of sputum could be a reflection of the microenvironment tumor. The secondary objective is to study the intestinal microbiota tract of patients receiving immunotherapy, depending on their consumption of antibiotics, and compare it to the pulmonary microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or over
* Diagnosis of metastatic NSCLC (Stage IV) adenocarcinoma only
* Absence of oncogenic addiction (EGFR, ALK, ROS1, RET, MET, BRAF)
* Treatment with ICI anti-PD1 or anti-PDL1 (pembrolizumab or atezolizumab) as 1st line treatment alone or in combination with chemotherapy and/or anti-angiogenic (bevacizumab).
* 1st injection of ICI, whether or not combined with chemotherapy

Exclusion Criteria:

* Patient under judicial protection
* Pregnant or breastfeeding women
* NSCLC of the epidermal or undifferentiated type
* Opposition to data processing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients suffering from adenocarcinoma type non-small cell lung cancer (NSCLC) without oncogenic addiction, metastatic, treated by ICI alone or in combination with 1st line chemotherapy at the Tours CHRU.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Immune and inflammatory response in the blood | 30 months
  * T cell sub populations assessed by their relative abundance, and will be expressed as a percentage of total T cells
  * B lymphocytes
  * Cytokine inflammatory profile: the level of activation/regulation, production of cytokines and cytotoxicity markers will be analysed as a percentage of cells expressing the markers or producing the cytokines in relation to the total cell population (e.g. HLA-DR+, CD38+, Bcl-2lo phenotype of CD8 T lymphocytes)
Immune and inflammatory response in the airways | 30 months
  * T cell sub populations assessed by their relative abundance, and will be expressed as a percentage of total T cells
  * B lymphocytes
  * Cytokine inflammatory profile: the level of activation/regulation, production of cytokines and cytotoxicity markers will be analysed as a percentage of cells expressing the markers or producing the cytokines in relation to the total cell population (e.g. HLA-DR+, CD38+, Bcl-2lo phenotype of CD8 T lymphocytes)

SECONDARY OUTCOMES:
Analysis of gut microbiota | 30 months
  characterisation of gut microbiota (16S rRNA sequencing)
Analysis of lung microbiota | 30 months
  characterisation of lung microbiota (16S rRNA sequencing)
perform blood pembrolizumab assays. | 30 months
  antibodies dosage
perform sputum pembrolizumab assays. | 30 months
  antibodies dosage

CONTACTS AND LOCATIONS:
Overall Officials: Marion FERREIRA, Principal Investigator — University Hospital, Tours
Locations (2):
- Ferreira Marion, Los Angeles, California, United States
- University hospital, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided